CLINICAL TRIAL: NCT06786442
Title: Clinical Efficacy Evaluation of a Skincare Product for Acne Face, Upper Chest and Back Used by Multiphototype Population Under Dermatological Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EV2309-0768 ZONIFICATION LABO
Record Dates: First submitted 2025-01-07; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Acne
Keywords: acne; truncal acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: all the three areas (face, upper chest, and back) need to conclude the study with a minimum of 75 valid cases (25 phototypes I-II / 25 phototypes III-IV / 25 phototypes V-VI. Mini 5 subjects per phototype).
Who Masked: Participant
Masking Description: Subjects will be identified by Screening Number (TXXX) and Inclusion/Randomization Number (R-00XX) at the very first study visit to maintain the confidentiality of their data.
  One hundred and thirty (130) subjects will be included to complete the study with at least seventy-five (75) valid cases for each assessment area, and among them:
  * 25 subjects with phototypes I and II for each assessment area;
  * 25 subjects with phototypes III and IV for each assessment area;
  * 25 subjects with phototypes V and VI for each assessment area.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FACE ACNE GROUP (Experimental): At least 75 subjects prone to acne of the face (25 phototypes I-II / 25 phototypes
  III-IV / 25 phototypes V-VI. Minimum 5 subjects per phototype):
  * Presenting at least 10 retentional lesions on the assessment zone
  * Presenting at least 5 inflammatory lesions on the assessment zone
  * Presenting at least 1 brown and/or red residual acne mark(s) on the assessment zone (the acne origin of these marks must be checked by the dermatologist by questioning the subject).
  EFFACLAR DUO+M CREAM application
  Interventions: Other: EFFACLAR DUO+M CREAM
- BACK ACNE GROUP (Experimental): At least 75 subjects prone to acne of the back (25 phototypes I-II / 25 phototypes
  III-IV / 25 phototypes V-VI. Minimum 5 subjects per phototype):
  * Presenting at least 10 retentional lesions on the assessment zone
  * Presenting at least 5 inflammatory lesions on the assessment zone
  * Presenting at least 1 brown and/or red residual acne mark(s) on the assessment zone (the acne origin of these marks must be checked by the dermatologist by questioning the subject).
  EFFACLAR DUO+M CREAM application
  Interventions: Other: EFFACLAR DUO+M CREAM
- UPPER CHEST ACNE GROUP (Experimental): At least 75 subjects prone to acne of the upper chest (25 phototypes I-II / 25 phototypes III-IV / 25 phototypes V-VI. Minimum 5 subjects per phototype): Presenting at least 10 retentional lesions on the assessment zone
  * Presenting at least 5 inflammatory lesions on the assessment zone
  * If possible (non-mandatory for this area): Presenting at least 1 brown and/or red residual acne mark(s) on the assessment zone (the acne origin of these marks must be checked by the dermatologist by questioning the subject).
  EFFACLAR DUO+M CREAM application
  Interventions: Other: EFFACLAR DUO+M CREAM

INTERVENTIONS:
Other: EFFACLAR DUO+M CREAM — twice a day: morning and evening. Subjects should be able to self-apply the product on all assessment areas (face, upper chest, and back)

SUMMARY:
The present aims to confirm, under normal conditions of use, the IP's clinical efficacy in controlling acne on the face, upper chest, and back after 28 and 42 days of product use, as well as illustrate its efficacy through standardized pictures. In addition, it is expected to assess the sensations of discomfort reported by participants at cutaneous levels, taking into consideration the product use guidelines determined by the manufacturer, and the self-perceived efficacy by participants immediately after the first application, after 7, 28, 42 days using the IP

DETAILED DESCRIPTION:
In accordance with ANVISA's definition on RDC 07 of 2015, personal hygiene products, cosmetics, and perfume are preparations composed of natural or synthetic substances, for external use on the various parts of the body such as skin, hair, nails, lips, external genital, teeth and mucous membranes of the oral cavity, with the exclusive or main purpose of cleaning and perfuming them, changing their appearance, correcting body odors, protecting and/or keeping them in good condition. It is of great importance that companies conduct clinical studies of their products so that consumers have maximum safety with the lowest risk of use. After confirming the evidence of safety of use by humans, the manufacturing company must submit the results obtained to ANVISA (whether the company intends to sell it in Brazil), as well as establishing label warnings and consumer service guidelines based on the information obtained. According to Helsinki Declaration and Brazilian legislation, any research involving human beings must comply with ethical premises. The purpose of them is to protect individuals' integrity, dignity, well-being, rights, and confidentiality. Therefore, studies involving personal care products, cosmetics and perfumes in safety investigation phase (i.e. investigational products) must follow the recommendations of Good Clinical Practices (GCP).

STATISTICAL ANALYSIS PLAN For each study assessment area (face, upper chest, and back), four statistical analysis will be conducted: one global analysis and one analysis per phototype cluster (I-II, III-IV, and V-VI). A total of 12 statistical analysis will be performed.

Parameters to be Analyzed:

* Number of papules;
* Number of pustules;
* Number of nodules;
* Number of blackheads;
* Number of microcysts;
* Number of excoriated lesions without inflammation;
* Number of red acne residual marks;
* Number of brown acne residual marks;
* Number of inflammatory lesions (papules + pustules + nodules). Calculated parameter
* Number of retentional lesions (blackhead + microcysts). Calculated parameter
* Number of acne residual marks (red acne residual marks + brown acne residual marks). Calculated parameter
* Number of other lesions (excoriated lesions without inflammation + residual marks).

Calculated parameter

▪ Total number of lesions (inflammatory lesions + total lesions + other lesions).

Calculated parameter

ELIGIBILITY:
Inclusion Criteria:

All phototypes - with at least 5 subjects of each phototype per assessment area:

* I, II: n=at least 25
* III, IV: n= at least 25
* V, VI: n=at least 25 All skin sensitivity (sensitive or non-sensitive); All skin types (dry, normal, combination or oily); Not presenting severe acne; All ethnicities; At least 75 subjects prone to acne of the face (25 phototypes I-II / 25 phototypes

III-IV / 25 phototypes V-VI. Minimum 5 subjects per phototype):

* Presenting at least 10 retentional lesions on the assessment zone
* Presenting at least 5 inflammatory lesions on the assessment zone
* Presenting at least 1 brown and/or red residual acne mark(s) on the assessment zone (the acne origin of these marks must be checked by the dermatologist by questioning the subject). At least 75 subjects prone to acne of the back (25 phototypes I-II / 25 phototypes

III-IV / 25 phototypes V-VI. Minimum 5 subjects per phototype):

* Presenting at least 10 retentional lesions on the assessment zone
* Presenting at least 5 inflammatory lesions on the assessment zone
* Presenting at least 1 brown and/or red residual acne mark(s) on the assessment zone (the acne origin of these marks must be checked by the dermatologist by questioning the subject). At least 75 subjects prone to acne of the upper chest (25 phototypes I-II / 25 phototypes III-IV / 25 phototypes V-VI. Minimum 5 subjects per phototype):
* Presenting at least 10 retentional lesions on the assessment zone
* Presenting at least 5 inflammatory lesions on the assessment zone
* If possible (non-mandatory for this area): Presenting at least 1 brown and/or red residual acne mark(s) on the assessment zone (the acne origin of these marks must be checked by the dermatologist by questioning the subject). Accepting to use their usual neutral sunscreen SPF (30 mini) daily and accepting not to expose themselves intensively to the sun and to use protection (hat and UV clothes, for example); Not presenting an excessive hair on the assessment areas; Not presenting tattoo in the assessment area that could interfere with the evaluations and with the possibility of exploiting the photographs; Able to apply the product to the whole application area;

Four weeks before study starts subject should:

* Not use any anti-acne/anti-sebum product;
* Use neutral cleanser;
* Use neutral sunscreen (minimum SPF 30);
* Not have exposed themselves intensively to the sun. Subjects in good general and mental health in the opinion of the investigator; Subjects demonstrating understanding of the study procedures, restrictions, schedule, and willingness to participate as evidenced by voluntary written informed consent. Subjects under 18 years old willing to participate will provide their written consent as well as their legal responsible.

Exclusion Criteria:

Pregnant or breastfeeding women; Any history of significant dermatological diseases or medical conditions may affect the clinical evaluation of the study product; Subjects currently using any medication, which in the opinion of the investigator, may affect the clinical evaluation of the study product; Previous history of atopy, allergic reactions, irritation, or intense discomfort feelings to similar products to the tested one; Visible sun-tanned skin; Subjects presenting excessive hair in the assessed areas (shaving of upper chest will only be accepted if already in the subject's usual routine for at least the last 3 months before inclusion visit); Having introduced new products within 4 weeks prior to the inclusion visit; Having performed any aesthetic procedures in the evaluated areas 12 months before study starts; Using any cosmetic products that may influence sebum control and/or claiming an action in the acne lesion or skin imperfections in the last month before study starts;

Previous aesthetic cares in the following periods before D0:

* Aesthetic procedures (chemical or mechanical peeling, dermabrasion, laser, pulsed light, etc.) on the evaluation areas - 12 months
* Oral retinoid-based treatment and injections on the evaluation areas- 6 months;
* Beginning, change or discontinuation of hormonal treatment (oestroprogesteron, cyproteron acetate, androgenic…) - 3 months;
* Cure of minerals or vitamin supplements (such as zinc, vitamin A, vitamin E…) - 3 months;
* Anti-acne and anti-seborrheic medical treatment (oral and topical), topical retinoid treatement and depigmenting/whitening product use - 2 months;
* Antibiotic and/or anti-inflammatory treatment (oral), aesthetic care at home or in a beauty salon (such as exfoliating scrub, mask) on the evaluation areas - 1 month;
* Exposure to direct sunlight or artificial UV, and self-tanning product on the evaluation areas - 1 month;
* Cosmetic products designated to regulate sebum secretion and/or acne - 1 month;
* Cosmetic products (skincare and/or make-up and/or shampoo) other than usual cleanser on the evaluation areas - 24 hours;
* Last shaving performed on the evaluation areas - 24 hours (men only); Having undergone aesthetics surgery on the evaluation areas; Permanent makeup: only on the lips and eyes are allowed, but without any retouching during the study; Having applied cosmetic products (skincare, make-up and/or cleanser) on the evaluation areas and/or shampoo and/or hairspray at day of inclusion visit;

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
Acne lesion and acne residual brown and red marks count | Day 0, Day 28 and Day 42
  The acne count will be performed based on the "LesionsCount Guidelines v 0.1" provided by the sponsor and acquired images will confirm the lesion location and accountability for all three areas. To assess the IP efficacy, at D0, D28 and D42, the dermatologist will perform an acne lesion and residual marks count by type as follows: inflammatory lesions (nodules, pustules and papules, including recently excoriated papules), non-inflammatory/retentional lesions (open comedones/blackheads, closed comedones/microcysts) and other lesions (excoriated lesions without inflammation and red acne residual marks and brown acne residual marks), for each assessment area (face, upper chest and back).

SECONDARY OUTCOMES:
Efficacy and Cosmetic acceptability through Self-assessment questionnaire | immediately after the first application (Day 0 T immediately), Day 7, Day 28 of product use and day 42 of product use
  To collect the participants' opinion and their perceptions regarding product efficacy
Illustrative photographies of tested areas | Day 0, Day 28 and Day 42
  Illustrative standardized images with Colorface device
Tolerance | Day 0, Day 28 and Day 42
  Safety feedback and report of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Thais Pontes, Dr, Principal Investigator — ARTHA
Locations (1):
- ARTHA, Rio de Janeiro, Centro Rj, Brazil

IPD SHARING:
Plan to Share IPD: No